CLINICAL TRIAL: NCT02758431
Title: Cardiovascular Consequences of Hypogonadism in Men
Brief Title: Cardiovascular Outcomes of Low Testosterone
Acronym: CardioVOLT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 15-1162; R01AG049762 (NIH)
Record Dates: First submitted 2016-04-20; First posted 2016-05-02 (Estimated); Last update posted 2024-10-10 (Actual); Status verified 2024-10

CONDITIONS: Hypogonadism
Keywords: testosterone
MeSH Terms: conditions — Hypogonadism | interventions — acyline; Anastrozole; Aromatase Inhibitors

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Group 1: Acyline plus placebo (No Testosterone Add-Back) (Placebo Comparator): Acyline plus placebo gel and placebo tablet.
  Interventions: Drug: Acyline; Drug: Placebo Gel; Drug: Placebo Tablet
- Group 2: Acyline plusTestosterone (Active Comparator): Acyline plus transdermal testosterone gel plus placebo tablet.
  Interventions: Drug: Acyline; Drug: Placebo Tablet; Drug: Testosterone Gel
- Group 3: Acyline plus Testosterone plus Arimidex) (Active Comparator): Acyline plus transdermal testosterone gel plus Aromatase inhibitor (Arimidex) oral.
  Interventions: Drug: Acyline; Drug: Testosterone Gel; Drug: Arimidex

INTERVENTIONS:
Drug: Acyline — Acyline 300ug/kg injection will be administered on Day 0 and on day 14
  Other Names: Gonadotropin releasing hormone antagonist
Drug: Placebo Gel — Placebo gel packet applied daily for 28 days.
  Other Names: Placebo
  Arms: Group 1: Acyline plus placebo (No Testosterone Add-Back)
Drug: Placebo Tablet — Placebo oral tablet taken daily for 28 days.
  Other Names: Placebo
  Arms: Group 1: Acyline plus placebo (No Testosterone Add-Back); Group 2: Acyline plusTestosterone
Drug: Testosterone Gel — Testosterone Gel applied daily for 28 days
  Other Names: Transdermal Testosterone Gel
  Arms: Group 2: Acyline plusTestosterone; Group 3: Acyline plus Testosterone plus Arimidex)
Drug: Arimidex — Arimidex Oral Tablet 1mg taken orally daily for 28 days
  Other Names: Aromatase inhibitor
  Arms: Group 3: Acyline plus Testosterone plus Arimidex)

SUMMARY:
This study plans to learn more about heart and vascular aging in men. In some men as they get older, testosterone levels fall below the normal range for young men. Also, as men get older cardiovascular health worsens. This can lead to high blood pressure and heart disease. In this study we want to find out what causes cardiovascular health to worsen in older men. Also we want to find out what happens when testosterone levels are lowered for a short time. Specifically, we want to see if the reduction in cardiovascular health in older men with low testosterone levels is because of damage to mitochondria. Mitochondria are the main power supply of the cells in our body. The results from this study will help to understand why cardiovascular health declines in older men with low testosterone levels compared to younger men and older men who have higher testosterone levels. Knowing this information will help to develop therapies to prevent heart disease in men.

DETAILED DESCRIPTION:
Cardiovascular (CV) aging, featuring large artery stiffening, endothelial dysfunction, and impaired left ventricular (LV) diastolic function, is a major risk factor for the development of cardiovascular diseases (CVD). Male aging is associated with a gradual and variable decline in serum testosterone (T) and low T is associated with accelerated CV aging. The purpose of this research is to determine the key functional mechanisms underlying accelerated CV aging in older men with low T. The overall hypothesis is that mitochondrial dysfunction and oxidative stress are mechanisms underlying the apparent accelerated CV aging in older men with low T. To test this hypothesis Aim 1 will use cross-sectional comparisons of young and older men with normal T (≥400 ng/dl), and older men with chronically low T (<300 ng/dl). To better isolate the effects of low T from factors that change with aging and chronic low T, Aim 2 will expand on the cross-sectional comparisons by assessing measures of CV function, oxidative stress burden and mitochondrial function in older men with normal T before and after randomization to short-term (28 d) gonadal suppression (gonadotropin releasing hormone antagonist, GnRHant) + placebo (PL), GnRHant+T alone, or GnRHant+T+aromatase inhibitor (AI). AI will control for the effects of aromatization of T to estradiol (E2), and thereby isolate T effects while suppressing E2, a potent modulator of CV function. The results from this research should provide new mechanistic insight into the processes that mediate the impairment in CV function at the cellular and systemic level in older men with low T. These studies will lead to a better understanding of the independent role of T in age-related changes in CV function and the mechanisms of action, which will help guide future sex-specific therapies for the prevention of CVD.

ELIGIBILITY:
Inclusion Criteria:

1. Men aged 18-40 years and 50-75 years
2. Chronically low testosterone group will have testosterone concentrations <300 ng/dl, and young and older normal testosterone groups will have testosterone levels 400-1000 ng/dl
3. No use of sex hormones for at least 1 year
4. Body mass index <40 kg/m2
5. Nonsmokers
6. Resting blood pressure <160/90 mmHg
7. Fasting plasma glucose <126 mg/dL
8. Healthy, as determined by medical history, physical examination, standard blood chemistries (chemistry panel, complete blood clot and circulating thyroid levels) and a graded exercise stress test with monitoring of blood pressure and electrocardiogram (ECG)
9. Sedentary or recreationally active (< 3 days/wk of vigorous aerobic exercise)
10. No use of medications that might influence cardiovascular function including anti-hypertensive, lipid lowering medications, and corticosteroids
11. No use of vitamin supplements or anti-inflammatory medications, or willing to stop 1 month prior and throughout the study.

Exclusion Criteria:

1. Contraindications to:

   1. Gonadotropin releasing hormone (GnRH) antagonist
   2. Testosterone gel and aromatase inhibitor including hypersensitivity to Acyline, Androgel®, Arimidex®
   3. Extrinsic peptide hormones, mannitol, GnRH or any other GnRH analogs
2. History of or active prostate or breast cancer or other sex hormone-dependent neoplasms
3. Pre-existing or active cardiac, renal or hepatic disease
4. History of stomach ulcer or bleeding
5. History of epilepsy or other seizure disorder
6. Diabetes
7. Active infection
8. Disease that affects the nervous system
9. Abnormal resting ECG

Additionally, men participating in the gonadal suppression intervention study will do so with the understanding that they will be randomly assigned to study groups that involve either GnRH antagonist plus testosterone gel plus placebo tablet (33% chance), GnRH antagonist plus testosterone gel plus aromatase inhibitor tablet (33% chance) or GnRH antagonist plus placebo gel plus placebo tablet (33% chance).

Ages: 18 Years to 75 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 232 (Actual)
Dates: Start 2016-07-01 (Actual); Primary Completion 2023-01-04 (Actual); Study Completion 2023-01-04 (Actual)

PRIMARY OUTCOMES:
Endothelial function | Change from baseline at 28 days
  Brachial artery flow-mediated dilation, and EndoPAT™
Carotid artery compliance | Change from baseline at 28 days
  Carotid artery compliance and beta stiffness index
Arterial stiffness | Change from baseline at 28 days
  Pulse-wave velocity
Left ventricular diastolic function | Change from baseline at 28 days
  Measured via Cardiac Echo

SECONDARY OUTCOMES:
NADPH oxidase | Change from baseline at 28 days
  Oxidative stress marker measured in endothelial cells
Nitrotyrosine | Change from baseline at 28 days
  Measured in endothelial cells
MnSOD | Change from baseline at 28 days
  Mitochondrial superoxide dismutase measured in endothelial cells
eNOS | Change from baseline at 28 days
  Endothelial nitric oxide synthase (eNOS) measured in endothelial cell
COX IV | Change from baseline at 28 days
  Marker of mitochondrial function measured in PBMCs
Mitochondrial RCR | Change from baseline at 28 days
  Mitochondrial respiration measured via Oroboros O2K

OTHER OUTCOMES:
Supine blood pressure | Change from baseline at 28 days
  On the cardiovascular testing days, supine blood pressure will be measured in triplicate.
Body Composition | Baseline
  Whole body and regional body composition will be determined using dual energy x-ray absorptiometry for subject characteristics and for the determination of fat-free mass for the AA dose preparation.
Plasma Lipid Concentrations | Baseline
  Plasma lipid concentrations, including total-cholesterol (C) and triglycerides (TG) will be determined at baseline. The rationale for making these measurements is for screening criteria, subject characteristics, and because they may correlate with CV function.
Glucose Concentrations | Change from baseline at 28 days
  Fasted glucose concentrations will be measured at screening and at each vascular test.
Sex Hormones | Change from baseline at 28 days
  Serum concentrations of total testosterone (T), estradiol, albumin, sex hormone binding globulin (SHBG), luteinizing hormone and follicle stimulating hormone will be measured to document changes in hormone concentrations and free T will be calculated using the known affinity constants of T for SHBG and for albumin. Additional measures of T will be measured after 60 days if testosterone has not returned to baseline. The 60 day plus measures are for safety.
Endothelin-1 (ET-1) | Change from baseline at 28 days
  Plasma ET-1 will be measured because it is a potent vasoconstrictor and has complex interactions with NO. Specifically, ET-1 synthesis is under tonic inhibition by NO.
Physical Activity Levels | Change from baseline at 28 days
  To document the habitual physical activity status at baseline and the last week of respective interventions, daily energy expenditure will be estimated using ActivPal monitors.

CONTACTS AND LOCATIONS:
Overall Officials: Kerrie Moreau, PhD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado CCTSI CTRC, Denver, Colorado, United States

IPD SHARING:
Plan to Share IPD: No